CLINICAL TRIAL: NCT03423693
Title: Comparative Study on Sputum Anti-inflammatory Mediators in Patients With Asthma or Asthma and COPD Overlap (ACOS) Syndrome, and COPD
Brief Title: Small Airway Obstruction in Asthma, COPD, ACOS
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Other Study IDs: Si527/2015
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Asthma; COPD; Asthma-COPD Overlap Syndrome
Keywords: Small airway obstruction; Asthma; COPD; ACOS
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sputum cell pellets, sputum supernatants, and sputum cytospins
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asthma with SAO+: Asthmatic patients with RV/TLC > or = 40
  Interventions: Other: No any intervention
- Asthma with SAO-: Asthmatic patients with RV/TLC < 40
  Interventions: Other: No any intervention
- ACO: Asthmatic patients with smoking > or = 10 pack years who have persistent airway obstruction (post-BD FEV1/FVC < 0.7) or COPD patients who have bronchodilator (BD) reversibility (absolute increase in FEV1 > or = 200 ml and FEV1% > or =12% after BD)
  Interventions: Other: No any intervention
- COPD: Patients with history of smoking > or = 10 pack year with post-BD FEV1/FVC < 0.7 and negative BD reversibility (absolute increase in FEV1 < 200 ml and FEV1% <12% after BD)
  Interventions: Other: No any intervention

INTERVENTIONS:
Other: No any intervention — No any intervention is applied to any groups in this study

SUMMARY:
This study was designed as retrospective chart review to test our hypothesis whether there are the differences in inflammatory and anti-inflammatory mediators between asthmatic and ACOS patients with small airway obstruction, and COPD

DETAILED DESCRIPTION:
The data including spirometry, lung volume, impulse oscillometry, sputum data, demographic characters within 6 months are collected for later analysis. Sputum supernatants and cytospins are used to determine inflammatory and anti-inflammatory responses in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma, ACO, and COPD
* Their spirometric, IOS, lung volume, demographic data and sputum samples are available

Exclusion Criteria:

* Concomitant diseases requiring immunosuppressive therapy
* Being on treatments with NSAIDs, macrolides, statins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited from Asthma Clinics and OPD in Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Lipoxin A4, , | 1 day (single time point)
  Lipoxin A4 is measured in sputum supernatants by ELISA

SECONDARY OUTCOMES:
IL-33 | 1 day (single time point)
  IL-33 is measured in sputum supernatants by ELISA
Thymic stromal lymphopoietin (TSLP) | 1 day (single time point)
  TSLP is measured in sputum supernatants by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong Maneechotesuwan, MD, PhD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No